CLINICAL TRIAL: NCT01795716
Title: Bioequivalence Study of Mesylate Imatinib Capsule in Chronic Myeloid Leukemia Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YMTN-1.0
Record Dates: First submitted 2013-02-06; First posted 2013-02-21 (Estimated); Results first posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mesylate imatinib capsule (Experimental): Single and multiple oral mesylate imatinib capsule 400mg qd
  Interventions: Drug: mesylate imatinib capsule
- Glivec (Active Comparator): Single and multiple oral Glivec 400mg qd
  Interventions: Drug: Glivec

INTERVENTIONS:
Drug: mesylate imatinib capsule — Single and multiple oral mesylate imatinib capsule 400mg qd
  Other Names: 111201
  Arms: mesylate imatinib capsule
Drug: Glivec — Single and multiple oral Glivec 400mg qd
  Other Names: Mesylate Imatinib tablet
  Arms: Glivec

SUMMARY:
1. purpose: To conduct the relative bioavailability study of a single dose and multiple doses of imatinib mesylate capsule (Jiangsu Chia-Tai Tianqing Pharmacy Co. Ltd.) versus Glivec (Novartis Pharma Stein AG).
2. Experimental Design： Two-period crossover design
3. Test drug: imatinib mesylate capsule Reference drug: Glivec
4. Sample size：20

DETAILED DESCRIPTION:
To conduct the relative bioavailability study of a single dose and multiple doses of imatinib mesylate capsule(Jiangsu Chia-Tai Tianqing Pharmacy Co. Ltd.) versus Glivec (Novartis Pharma Stein AG) and compare the bioequivalence and pharmacokinetics of the two products in 20 patients with chronic myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic myeloid leukemia;
* Age: 18-65 years,gender:both.
* Weight: standard weight ± 20% within, and avoid weight disparity is too large;
* No previous radiation therapy, chemotherapy, or surgery within 1 weeks before treatment with imatinib;
* Performance status 0 to 3 (WHO scale); Life expectancy greater than 3 months;
* No other malignancy;
* Adequate hepatic, renal, and bone marrow function (WBC≥3.0×109/L，ANC≥1.5×109/L，PLT≥80×109/L. Serum bilirubin≤1.5×the institutional upper limit of normal, ALT、ALP≤2.5×the institutional upper limit of normal, creatinine≤1.5×the institutional upper limit of normal);
* Ability to understand objectives of the study, the study procedure, the pharmacological properties of the drug and possible adverse reactions and the willingness to sign a written informed consent.

Exclusion Criteria:

* Suffering from heart, liver, kidney disease or severe acute and chronic gastrointestinal diseases;
* Pregnant or lactating women and be sensitive to drug;
* Subjects are thought unsuitable for the study by investigators;
* Inability to comply with protocol or study procedures in the opinion of the investigator;
* Attending other clinical trials or attended other clinical trials 3 months ago.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shen Zh xiang, doctor, Principal Investigator — Shanghai Jiaotong University School of Medicine Ruijin Hospital
Locations (1):
- Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesylate Imatinib Capsule First, Then Glivec: Eligible subjects were randomly assigned to receive a single and multiple 400 mg oral dose Mesylate Imatinib Capsule during the first study period.In the first phase of the multiple-dose administration, the groups were given Mesylate Imatinib Capsule 400 mg once daily in the morning for ten consecutive days. After ten-day washout period, then Glivec was administered under the same protocol .
- Glivec First, Then Mesylate Imatinib Capsule: Eligible subjects were randomly assigned to receive a single and multiple 400 mg oral dose Glivec during the first study period. In the first phase of the multiple-dose administration, the groups were given Glivec 400 mg once daily in the morning for ten consecutive days. After ten-day washout period, then Mesylate Imatinib Capsule was administered under the same protocol .
Period: First Intervention (13 Days)
Arm/Group | Mesylate Imatinib Capsule First, Then Glivec | Glivec First, Then Mesylate Imatinib Capsule
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0
Period: Washout (10 Days)
Arm/Group | Mesylate Imatinib Capsule First, Then Glivec | Glivec First, Then Mesylate Imatinib Capsule
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0
Period: Second Intervention (13 Days)
Arm/Group | Mesylate Imatinib Capsule First, Then Glivec | Glivec First, Then Mesylate Imatinib Capsule
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mesylate Imatinib Capsule First, Then Glivec: Eligible subjects were randomly assigned to receive a single and multiple 400 mg oral dose Mesylate Imatinib Capsule during the first study period. In the first phase of the multiple-dose administration, the groups were given Mesylate Imatinib Capsule 400 mg once daily in the morning for ten consecutive days. After ten-day washout period, then Glivec was administered under the same protocol .
- Total: Total of all reporting groups
Arm/Group | Mesylate Imatinib Capsule First, Then Glivec | Glivec First, Then Mesylate Imatinib Capsule | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Geometric Mean (Full Range); unit: years] | 33 [17 to 59] | 33 [17 to 59] | 33 [17 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  China | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Area Under Curve (AUC) Time Frame: Predose, 0.5,1,1.5,2,3,5,8,12,24,48,72hours Post-dose
Time Frame: predose, 0.5,1,1.5,2,3,5,8,12,24,48,72hours post-dose
Measure: Mean (Standard Deviation); unit: mcg*hr/mL
Groups:
- Mesylate Imatinib Capsule: Eligible subjects were assigned to receive a single and multiple 400 mg oral dose Mesylate Imatinib Capsule
- Glivec: Eligible subjects were assigned to receive a single and multiple 400 mg oral dose Glivec
Arm/Group | Mesylate Imatinib Capsule | Glivec
Number analyzed (Participants) | 21 | 21
mcg*hr/mL | 37256 (11442) | 37206 (10620)
Statistical Analysis 1: Comparison: Mesylate Imatinib Capsule vs Glivec; The 90% confidence intervals of the test/reference ratios for AUC0-∞ and Cmax were determined. Log-transformed data were used in the analysis. Following international guidelines (including those of the SFDA), the test and reference for mutations were considered bioequivalent if the 90% CIs of the test/reference ratios of AUC was within range of 0.80 to 1.25 and Cmax was within 0.70 to 1.43; Test type: Non-Inferiority or Equivalence — The 90%CIs of the test/reference ratios for AUC0-∞ and Cmax were determined. Log-transformed data were used in the analysis. Following international guidelines (including those of the SFDA), the test and reference for mutations were considered bioequivalent if the 90% CIs of the test/reference ratios of AUC was within range of 0.80 to 1.25 and Cmax was within 0.70 to 1.43; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 29 days
Groups:
- Mesylate Imatinib Capsule: Subjects were assigned to receive a single and multiple 400 mg oral dose Mesylate Imatinib Capsule
- Glivec: Subjects were assigned to receive a single and multiple 400 mg oral dose Glivec
Arm/Group | Mesylate Imatinib Capsule | Glivec
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 10/21 | 13/21
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesylate Imatinib Capsule (N=21) | Glivec (N=21)
nausea and vomit (Gastrointestinal disorders) | 10 (10) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No